CLINICAL TRIAL: NCT03845543
Title: Belgian-Italian Prospective, Single Arm, Multicentre Study to Evaluate the Efficacy and Safety of BTK Treatment With the Luminor 14 Paclitaxel Coated Percutaneous Transluminal Angioplasty Balloon Catheter of iVascular of 150 Subjects With Critical Limb Ischemia
Brief Title: Belgian-Italian Trial to Evaluate the Efficacy and Safety of Below The Knee (BTK) Treatment With the Luminor 14 Paclitaxel Coated Percutaneous Transluminal Angioplasty Balloon Catheter of iVascular
Acronym: BIBLIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBLIOS-Luminor14BTK
Record Dates: First submitted 2019-01-09; First posted 2019-02-19 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luminor-14 paclitaxel eluting balloon (Experimental): Pre-dilatation of 180 seconds with a standard non-drug-coated semi-compliant balloon followed by a dilatation with a Luminor-14 paclitaxel eluting balloon (3µg/mm² balloon surface).
  Interventions: Device: Luminor-14 Paclitaxel eluting balloon

INTERVENTIONS:
Device: Luminor-14 Paclitaxel eluting balloon — Patients will be treated with the Luminor-14 paclitaxel eluting balloon

SUMMARY:
The BIBLIOS trial investigates the efficacy and safety of BTK treatment of patients suffering from critical limb ischemia (Rutherford 5) with the Luminor-14 Paclitaxel coated Percutaneous Transluminal Angioplasty Balloon catheter of iVascular. An expected total of 150 patients will be treated. Infrapopliteal lesions will be treated during this trial. The Paclitaxel eluting balloon Luminor-14 is designed for percutaneous transluminal angioplasties in which the balloon will dilate the artery upon inflation. The balloon is coated with Paclitaxel intended to avoid cellular proliferation. The drug is released by means of rapid inflation as to release a high dose in a short amount of time. Patients will be invited for a follow-up visit at 1, 6 and 12 months post-procedure. The primary efficacy endpoint is defined as freedom from major adverse limb events, defined as above the ankle target limb amputations or major reintervention to the target lesions at 6 months. The primary safety endpoint is freedom from major adverse limb event at 30 days. The secondary endpoints consist of functional flow in target vessel, freedom from clinically driven target lesion revascularisation, above the ankle amputation free survival and limb salvage at 6 and 12 months, and also procedural success, wound healing status and wound healing time.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to assess the safety and efficacy of the Luminor-14 DCB for the treatment of infrapopliteal lesions patients with critical limb ischemia.

The patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should be geographically stable, willing and able to cooperate in this clinical study, and remain available for long term follow-up. The patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following will be collected: an informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of acute limb ischemia (Rutherford category), the resting ankle-brachial index (ABI), life quality and if applicable a wound assessment.

During the procedure the guidewire will cross the entire study lesion after which the lesion will be assessed through angiography. A pre-dilatation with a standard non-drug-coated balloon will be performed followed by a dilatation of the lesion with a Luminor-14 balloon (iVascular). If dilatation was not successful (>30% stenosis, perforation, occlusive or flow limiting dissection) prolonged inflation should be attempted after which bail-out stenting with a non-drug-coated dedicated BTK stent is allowed in case of inadequate results.

The regular follow-up is necessary to monitor the condition of the patient and the results of the procedure. Patients will be invited on weekly follow-up, with special attention to wound healing status at each visit until the wound is completely healed. The other required follow-up visits are 1,6 and 12 months follow-ups. During these visit the following data will be collected: medication record, physical exam, wound assessment and healing status, quality of life, duplex ultrasound of target vessel and possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females ≥ 18 years of age at the time of consent. Females of childbearing potential have a negative pregnancy test <7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation. Female participants will be exempted from this requirement in case they are sterile, infertile or have been post-menopausal for at least 12 months
* Subject has been informed of and understands the nature of the study and provides signed informed consent to participate in the study. If the subject possesses the ability to understand and provide informed consent but due to physical inability, the subject cannot sign the informed consent form. An impartial witness may sign on behalf of the subject.
* Willing to comply with all required follow-up visits
* Rutherford Classification 5
* Significant degree of stenosis >70% or chronic total occlusion (CTO)
* Infrapopliteal lesion: P3 to the ankle-joint level (not below-the-ankle (BTA)); full length lesions or tandem lesions are allowed
* Wound, Ischemia, foot Infection (WIfI) tissue loss grade 1-2 at baseline
* WIfI foot infection grade of 0-2 at baseline
* WIfI ischemia grade 2-3 at baseline
* Estimated life expectancy ≥ 1 year
* Multiple lesions can be treated if they are located in separate vessels per standard of care but only one (1) BTK vessel can be considered as the target lesion/vessel and need to be treated according the Clinical Investigation Protocol (CIP) guidelines.
* Target vessel should give direct or indirect run-off to the foot (clearly documented in a foot/BTA angiogram)
* Patients with in-flow lesions can be included if the lesions are treated successfully (residual stenosis ≤30%) with the same drug coated balloon (DCB) platform, bail-out stenting with a bare-metal stent (BMS).
* Successful pre-dilatation of the target lesion (≤30% residual stenosis)

Exclusion Criteria:

* Previous bypass graft in the target limb
* Acute limb ischemia, defined as symptom onset during less than 14 days prior to the index procedure
* Prior or planned above-the-ankle amputation to the target limb (this does not apply to ray amputation of ≤2 digits, simple digital amputations or ulcer debridement)
* Previous DCB treatment in target vessel 6 months prior to index procedure
* WIfI tissue loss grade 0 or 3 at baseline
* WIfI foot infection grade 3 at baseline
* WIfI ischemia grade 0-1 at baseline
* Any systemic infection or immunocompromised state. Patients with an ascending infection/deep foot infection or abscess/white blood count (WBC)≥12.000/or febrile state or C reactive protein (CRP)>5mg/L
* Endovascular or surgical procedure (not including diagnostic procedures, planned simple digital amputation or wound debridement) to the target limb within 30 days after the index procedure
* Existing stent implant in the target vessel
* Use of alternative therapies: atherectomy, cutting/scoring balloons, laser, …
* Known coagulopathy, hypercoagulable state, bleeding diathesis, other blood disorder, or a platelet count less than 80.000/μL or greater than 500.000/μL
* Any subject in which antiplatelet, anticoagulant or thrombolytic therapy is contraindicated
* Myocardial infarction, coronary thrombolysis or angina less than 30 days prior to the index procedure
* History of stroke or transient ischemic attack (TIA) less than 90 days prior to the index procedure
* Known hypersensitivity or contraindication to nickel-titanium alloy (Nitinol)
* Has other comorbidities that, in the opinion of the investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up
* Patients on haemodialysis
* Known hypersensitivity or allergy to contrast agents that cannot be medically managed
* Known hypersensitivity or allergy to heparin, aspirin, paclitaxel, clopidogrel or other antiplatelet/anticoagulant therapies
* Inadequate inflow lesion treatment (>30% residual stenosis)
* Inadequate result of pre-dilatation (>30% residual stenosis)
* Inadequate run-off to the foot
* Bilateral BTK enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Study Director — ID3 Medical
Locations (9):
- Belgium (6):
  - OLV Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk
  - AZ Groeninge, Kortrijk
  - Regionaal Ziekenhuis Heilig Hart, Tienen
- Italy (2):
  - Policlinico Abano Terme, Abano Terme, Padua
  - IRCCS Policlinico San Donato, San Donato
- Hospital Univ. Germans Trias I Pujol, Badalona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Started | 150
Completed | 94
Not Completed | 56
Not completed — Death | 25
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 12
Not completed — Adverse Event | 17

BASELINE CHARACTERISTICS:
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 131
  Italy | 9
  Spain | 10
Nicotine abuse [Count of Participants; unit: Participants] | 53
Hypertension [Count of Participants; unit: Participants] | 120
Hypercholesterolemia [Count of Participants; unit: Participants] | 99
Previous arterial intervention [Count of Participants; unit: Participants] | 73
Previous coronary intervention [Count of Participants; unit: Participants] | 51
Previous cerebrovascular interventions [Count of Participants; unit: Participants] | 6
Diabetes [Count of Participants; unit: Participants] | 107
Obesity [Count of Participants; unit: Participants] | 41
Renal insufficiency [Count of Participants; unit: Participants] | 52

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Freedom From MALE
Description: Freedom from major adverse limb events (MALE) defined as absence of above-ankle target limb amputation or major re-intervention to the target lesion(s) (i.e. new bypass graft, jump/interposition graft revision or thrombectomy/thrombolysis).
Time Frame: 6 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants | 144

2. Primary Outcome: Primary Safety Endpoint: Freedom From MALE
Description: Freedom from major adverse limb events defined as absence of above-ankle target limb amputation or major re-intervention to the target lesion(s) (i.e. new bypass graft, jump/interposition graft revision or thrombectomy/thrombolysis).
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants | 148

3. Primary Outcome: Primary Safety Endpoint: Freedom From POD
Description: No peri-operative death (POD) related to device, procedure or any other cause.
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants | 146

4. Secondary Outcome: Target Vessel Functional Flow Assessment
Description: Target vessel functional flow assessment defined as the presence of blood flow using duplex ultrasound. Evidence of no blood flow within the treated segment indicates loss of patency.
Time Frame: 6 and 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants
  6 months | 133
  12 months | 129

5. Secondary Outcome: Freedom From Clinically Driven Target Vessel Revascularisation
Description: Freedom from clinical driven target lesion revascularization defined as absence of any reintervention due to clinical deterioration, defined as a worsening of the patient's quality of life, reflected by the health-questionnaire (EQ-5D), worsening of the Rutherford category with minimal 1 class or worsening of wound status.
Time Frame: 6 and 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants
  6 months | 138
  12 months | 133

6. Secondary Outcome: Amputation Free Survival
Description: Amputation free survival defined as alive with freedom from any above the ankle target limb amputation
Time Frame: 6 and 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants
  6 months | 130
  12 months | 119

7. Secondary Outcome: Limb Salvage
Description: Limb salvage is defined as freedom from any above the ankle target limb amputation
Time Frame: 6 and 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants
  6 months | 144
  12 months | 143

8. Secondary Outcome: Procedural Success
Description: Procedural success is defined as restoration of at least 1 below the knee artery with <30% residual stenosis in the final angiogram and outflow into the foot.
Time Frame: During index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
Participants | 142

9. Secondary Outcome: Mean Wound Healing Status
Description: At 1, 6 and 12 months visits, the healing status of each wound will be scored based on 3 parameters:
  Wound's diameter: 0 points for wounds with diameter >9cm², 1 point for wounds with diameter 1-9cm², 2 points for wounds with diameter <1cm² Wound's depth: 0 points for depth to the bone/joint wounds, 1 point depth to muscle/tendon wounds, 2 points depth to the skin or subcutaneous wounds
  % granulation tissue: 0 points for a wound with <50% red granulation tissue, 1 point for a wound with 50-75% red granulation tissue, 2 points for a wound with >75% red granulation tissue A total wound healing score is calculated by combining the 3 parameter points. E.g.:wound with diameter 1-9cm², depth to the bone, and <50% red granulation tissue has a score of 1+0+0=1. A wound with a score 6/6 is the best possible score for a non-healed wound while a 0/6 is the worst score a wound can have.
  After all total wound healing scores are calculated, a mean for each follow-up visit is calculated.
Time Frame: 1, 6 and 12 months post-procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
score on a scale
  1 month | 4.4 (1.4)
  6 months | 4.4 (1.4)
  12 months | 4 (1.3)

10. Secondary Outcome: Wound Healing Time
Description: Wound healing time is defined as the number of days needed for the wound to heal completely after the index procedure.
Time Frame: 1, 6 and 12 months post-procedure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
Number analyzed (Participants) | 150
days | 144 (103)

ADVERSE EVENTS:
Time Frame: 12 months post-procedure
Arm/Group | Luminor-14 Paclitaxel Eluting Balloon
All-Cause Mortality (participants affected / at risk) | 25/150
Serious Adverse Events (participants affected / at risk) | 88/150
Other Adverse Events (participants affected / at risk) | 45/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luminor-14 Paclitaxel Eluting Balloon (N=150)
Anemia (Blood and lymphatic system disorders) | 4 (7)
Cerebro vascular incident (Blood and lymphatic system disorders) | 1 (1)
Septic shock resulted in death (Blood and lymphatic system disorders) | 1 (1)
Shock (Blood and lymphatic system disorders) | 1 (1)
Arrhythmias (Cardiac disorders) | 2 (2)
CVA resulted in death (Blood and lymphatic system disorders) | 1 (1)
Heart disorder resulted in death (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 3 (3)
Reticulopathy (Eye disorders) | 1 (1)
Cancer resulted in death (Gastrointestinal disorders) | 1 (1)
Stomach ulcer (Gastrointestinal disorders) | 2 (2)
Other (Gastrointestinal disorders) | 2 (2)
Deterioration of general health (General disorders) | 2 (2)
Detoriation of general health resulted in death (General disorders) | 11 (11)
Other (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Covid infection resulted in death (Infections and infestations) | 4 (4)
Infected foot wound (Infections and infestations) | 9 (9)
Lung infection resulted in death (Infections and infestations) | 2 (2)
Other (Infections and infestations) | 4 (4)
Accidental fall (Injury, poisoning and procedural complications) | 5 (5)
Accidental fall resulted in death (Injury, poisoning and procedural complications) | 2 (2)
Foot wound (Musculoskeletal and connective tissue disorders) | 2 (2) — Foot wound with bone contact or amputation
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 10 (10)
Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Other (Nervous system disorders) | 2 (2)
Gallstone (Renal and urinary disorders) | 2 (2)
Kidney failure (Renal and urinary disorders) | 2 (4)
Kindey faillure resulted in death (Renal and urinary disorders) | 1 (1)
Other (Renal and urinary disorders) | 1 (1)
Breast cancer (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial stenosis/occlusion (Vascular disorders) | 34 (53)
Other (Vascular disorders) | 5 (5)
Foot wound (Skin and subcutaneous tissue disorders) | 24 (32)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luminor-14 Paclitaxel Eluting Balloon (N=150)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Other (Cardiac disorders) | 2 (2) — Arrhytmia, cardiomyopathy
Dental removal (Gastrointestinal disorders) | 1 (1)
Deterioration of general health (General disorders) | 2 (2)
Other (General disorders) | 1 (1)
Skin irritation (Immune system disorders) | 1 (1)
Foot wound (Infections and infestations) | 4 (4)
Other (Infections and infestations) | 2 (2)
Accidental fall (Infections and infestations) | 3 (3)
Other (Musculoskeletal and connective tissue disorders) | 4 (5)
Kidney faillure (Renal and urinary disorders) | 1 (1) — Worsening of chronic kidney failure
Other (Renal and urinary disorders) | 2 (2)
Foot wound (Skin and subcutaneous tissue disorders) | 17 (24)
Pseudoaneurysm (Vascular disorders) | 4 (4)
Arterial stenosis/occlusion (Vascular disorders) | 8 (8)
Dissection (Vascular disorders) | 2 (2)
Other (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to make announcements or oral presentations in any context without the Sponsor's prior written consent, except as required by law or by court administrative order. The relevant manuscripts shall be thus submitted to the Sponsor for approval to ensure that no confidential matters are made public. Once clinical research and/or results have been approved for publication by the Sponsor, they are no longer subjected to this provision in regards to any form of disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03845543/Prot_SAP_000.pdf